CLINICAL TRIAL: NCT00043095
Title: A Phase I Trial of BMS 247550 (NSC# 710428) and Gemcitabine in Patients With Advanced Solid Tumor Malignancies
Brief Title: BMS-247550 and Gemcitabine in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000256333; MSKCC-02012; NCI-5696
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2005-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Gemcitabine; ixabepilone

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining BMS-247550 with gemcitabine in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose, dose-limiting toxicity, and safety of BMS-247550 when combined with gemcitabine in patients with advanced solid tumors.
* Determine the plasma pharmacokinetics of this regimen in this patient population.
* Assess, preliminarily, any antitumor activity of this regimen in this patient population.

OUTLINE: This is a dose-escalation study of BMS-247550.

Patients receive gemcitabine IV over 90 minutes on days 1 and 8 followed by BMS-247550 IV over 3 hours on day 8. The order of chemotherapy drug administration on day 8 is reversed during the second course only. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BMS-247550 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 9 patients total are treated at the MTD.

PROJECTED ACCRUAL: A maximum of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-hematological cancer that is unresponsive to currently available therapies or for which there is no known effective treatment
* Clinical or radiological evidence of disease required
* No active brain metastases, including evidence of cerebral edema (by CT scan or MRI), progression from prior imaging study, any requirement for steroids, or clinical symptoms

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin at least 8.0 g/dL

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* ALT and AST no greater than 2.5 times upper limit of normal (ULN) or 93 U/L

Renal

* Creatinine no greater than 1.5 times ULN or 2.0 mg/dL

Other

* No documented hypersensitivity reaction to prior paclitaxel or other therapy containing Cremophor EL
* No grade 2 or greater pre-existing peripheral neuropathy
* No serious uncontrolled medical disorder or active infection that would preclude study therapy
* No dementia or altered mental status that would preclude informed consent
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior immunotherapy

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin, or doxorubicin HCl liposome)
* Prior taxanes allowed
* Prior adjuvant or neoadjuvant chemotherapy allowed
* No more than 2 prior chemotherapy regimens in the metastatic setting
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent hormonal therapy except hormone-replacement therapy
* Concurrent medications to maintain castrate status for progressive hormone-refractory prostate cancer allowed

Radiotherapy

* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow
* No concurrent radiotherapy

Surgery

* Not specified

Other

* At least 4 weeks since prior investigational agents
* No other concurrent experimental anticancer medications
* No concurrent alternative therapies (e.g., high-dose vitamins or herbal medicines)
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-06

CONTACTS AND LOCATIONS:
Overall Officials: Sibyl Anderson, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States